CLINICAL TRIAL: NCT02487680
Title: Effect of a Table Water Enriched With Amino Acids and Chromium on Blood Glucose and Insulin Levels After a Meal
Brief Title: Effects of an Amino Acid and Chromium-picolinate Containing Drink on Glucose Metabolism on Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DoubleGood AB (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: DoubleGood Lund
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breakfast meal (Experimental): A breakfast like meal will be provided together with a drink to overnight fasted subjects
  Interventions: Dietary Supplement: Amino Acids and chromium-picolinate containing drink; Dietary Supplement: Placebo drink
- Lunch meal (Experimental): A lunch like meal will be provided together with a drink to overnight fasted subjects
  Interventions: Dietary Supplement: Amino Acids and chromium-picolinate containing drink; Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Amino Acids and chromium-picolinate containing drink — Evaluation of the dietary supplement drink containing amino acids and chromium picolinate and aroma
Dietary Supplement: Placebo drink — Evaluation of the placebo supplement drink containing only aroma

SUMMARY:
It has previously been shown in healthy overweight subjects, that table water including a defined amount of amino acids and chromium can decrease the postprandial glucose. In this study, the effect of this table water on glucose excursions after a test meal containing a defined amount of available carbohydrates, protein and fat will be studied in healthy subjects. The study will be conducted in a cross -over design, double blinded and placebo controlled including 20 participants. The primary endpoint of the study is the incremental area under the curve for plasma glucose (iAUCgluc) within 180 minutes after ingestion of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Stable body weight (no changes above 3 kg during the last 2 months)
* Good general health
* Body mass index 19 - 30 kg/m2 (normal to overweight)
* Fasting blood glucose below 6.1 mmol/L

Exclusion Criteria:

* Any medication that could influence the study. Such as medication against diabetes, hypoglycemia, hypertension or hypercholesterolemia
* Psychiatric Disease
* Alcohol or drug abuse
* Smokers or people consuming snus
* Acute infections
* Vegetarians/vegans
* Suffering from Lactose or Gluten intolerance
* Pregnancy or Lactation
* Participation in another study at the same time
* Any other parameter that the PI will judge as inadequate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve for Glucose after ingestion of a test meal | 180 min

SECONDARY OUTCOMES:
Area under the curve for insulin after ingestion of a test meal | 180 min

CONTACTS AND LOCATIONS:
Overall Officials: Per Humpert, MD, Prof, Principal Investigator — Stoffwechselzentrum Rhein Pfalts, Mannheim, Germany and Department of internal medicine, University of Heidelberg, Germany; Ana Rascón, PhD, Prof, Study Director — Food for Health Science Center, Lund University, Sweden; Kristina Andersson, PhD, Study Chair — Experimental Medical Science, Lund University, Sweden